CLINICAL TRIAL: NCT01596608
Title: Efficacy and Tolerability of Magnetic Seizure Therapy (MST) as an Alternative to Electroconvulsive Therapy (ECT) for Treatment Resistant Depression, Schizophrenia, and Obsessive Compulsive Disorder
Brief Title: Magnetic Seizure Therapy (MST) for Treatment Resistant Depression, Schizophrenia, and Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Z. J. Daskalakis, Chair, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 145-2010
Record Dates: First submitted 2012-05-08; First posted 2012-05-11 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Depressive Disorder; Schizophrenia; Schizoaffective Disorder; Obsessive-Compulsive Disorder
Keywords: Magnetic seizure therapy; Treatment resistance; Open-label trial; Treatment resistant depression; Treatment resistant schizophrenia; Treatment resistant obsessive-compulsive disorder
MeSH Terms: conditions — Depressive Disorder; Schizophrenia; Psychotic Disorders; Obsessive-Compulsive Disorder; Depressive Disorder, Treatment-Resistant; Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magnetic Seizure Therapy (Experimental)
  Interventions: Device: Magnetic Seizure Therapy (MagPro MST)

INTERVENTIONS:
Device: Magnetic Seizure Therapy (MagPro MST) — 100% machine output at between 25 and 100 Hz, with coil directed over frontal or vertex brain regions, until adequate seizure achieved. Six treatment sessions, at a frequency of two or three times per week will be administered. If subjects fail to achieve the pre-defined criteria of remission at that point, the dose will be increased to the maximal stimulator output and 3 additional treatment sessions will be provided. This will be repeated a total of 5 times (i.e., maximum treatment number is 24). 24 treatments is typically longer that a conventional ECT treatment course. However, evidence does suggest that longer treatment courses may be needed with MST, particularly in more treatment resistant psychiatric conditions such as OCD and schizophrenia.
  Other Names: MagPro MST (Tonica Elektronik A/S, Denmark)

SUMMARY:
Electroconvulsive therapy (ECT) has unparalleled efficacy in treating severe depression, and is also useful in treatment-refractory cases of schizophrenia and obsessive compulsive disorder (OCD). However, its use is limited by significant adverse effects on memory and cognition. In addition, ECT cannot be precisely targeted, since it relies on unpredictable pathways of electrical conduction through the brain. Magnetic seizure therapy (MST) is currently under investigation as a targetable, cognition-sparing alternative to ECT. MST uses magnetic fields rather than electrical stimuli for seizure induction, dramatically reducing the passage of induced current through undesired brain regions. 10 years of experimental studies have established the safety of MST in animal and human subjects. This pilot study will investigate whether MST has similar efficacy to ECT, with fewer cognitive side effects, in patients with severe depression, schizophrenia, and OCD.

DETAILED DESCRIPTION:
Although ECT is effective against severe depression, psychosis, and OCD, it also produces significant impairments of autobiographical memory and other cognitive functions. These side effects limit the acceptability and tolerability of ECT in many patient populations. They also limit the number of treatments that can be administered in a course of ECT, leading to high relapse rates once ECT is discontinued. In animal studies, MST has been shown to have far fewer adverse cognitive effects than ECT. In small human studies, humans have shown faster subjective and objective recovery of orientation after MST than with ECT. However, the precise degree of cognitive sparing in MST versus ECT has yet to be established. Likewise, the comparative efficacy of MST versus ECT in severe depression, schizophrenia, and OCD remains to be seen. The investigators aim to determine whether MST spares autobiographical memory and other cognitive functions, while retaining comparable efficacy to that of ECT.

Objective 1: To compare the efficacy of MST and ECT in treating patients with severe depression, schizophrenia, and OCD.

Hypothesis 1: MST will have equivalent efficacy to ECT on objective measures of mood, schizophrenia, and OCD symptoms.

Objective 2: To compare the effects of MST and ECT on autobiographical memory and other cognitive functions in patients with severe depression, schizophrenia, schizoaffective disorder and OCD.

Hypothesis 2: MST will have significantly lower adverse effects on objective measures of autobiographical memory and other cognitive functions in patients with severe depression, schizophrenia, and OCD.

Objective 3: To compare the changes in brain function that result from MST and ECT.

Hypothesis 3: Both MST and ECT will produce changes in functional brain activity consistent with antidepressant response, antipsychotic response, and antiobsessive response, along with a sparing of cognitive functions.

The discovery of a viable alternative to ECT, with equivalent efficacy but fewer side effects, would have a transformative effect on the treatment of several forms of severe mental illness. At present, many patients who could benefit from ECT do not pursue this treatment due to concerns about cognitive side effects, as well as the enduring social stigma of ECT itself. In addition, many patients who have benefited from ECT are obliged to discontinue this effective treatment because of mounting cognitive side effects; high rates of relapse then ensue.

If MST could be shown to spare autobiographical memory and other forms of cognition, many more patients would be willing to take advantage of the treatment. They would also be able to continue the treatment, when effective, for longer periods. The potential result would be a dramatic improvement in the rates of remission and relapse for patients with severe depression and other forms of mental illness.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 to 85
* DSM-IV diagnosis of major depressive episode with or without psychotic features in the context of MDD or bipolar disorder; OCD or Schizophrenia
* 24-item HRSD score of ≥ 21 (for depression subjects)
* 18-item BPRS score of ≥ 37 (for schizophrenia subjects)
* Y-BOCS score of ≥ 16 (for OCD subjects)
* demonstrate capacity to give informed consent
* are a Canadian resident

Exclusion Criteria:

* have an unstable medical and/or neurological condition
* are currently pregnant or lactating
* are not considered sufficiently well to undergo general anesthesia for any reason
* have a cardiac pacemaker, cochlear implant, implanted electronic device or non-electric metallic implant
* are taking a benzodiazepine at a dose greater than lorazepam 2mg or equivalent
* are taking any non-benzodiazepine anticonvulsant
* have active substance misuse or dependence within the past 3 months
* have a current diagnosis of delirium, dementia or another cognitive disorder secondary to a general medical condition
* have a co-morbid borderline personality disorder and/or antisocial personality disorder
* have had a history of any suicide attempts in the past 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Score on rating scale that corresponds to diagnosis: i) Hamilton Rating Scale for Depression, 24-item (HRSD-24); or ii) Yale-Brown Obsessive Compulsive Scale (Y-BOCS); or iii) Brief Psychiatric Rating Scale (BPRS) | Change from baseline in HRSD-24 / Y-BOCS / BPRS at date of symptom remission or date of the 24th treatment, whichever comes first, assessed up to 12 weeks
  i) The HRSD-24 is a semi-structured, clinician-administered scale used to assessed the severity of depressive symptoms.
  ii) The Y-BOCS is a clinician-rated scale used to assess the severity of OCD symptoms.
  iii) The BPRS is a clinician-administered scale used to assess the severity of various psychiatric symptoms, such as depression, anxiety, hallucinations, and delusions. In this study, it will be used with participants diagnosed with schizophrenia.
Score on rating scale that corresponds to diagnosis: i) HRSD-24; or ii) Y-BOCS; or iii) BPRS | Change from baseline in HRSD-24 / Y-BOCS / BPRS at 1 month after final treatment
Score on rating scale that corresponds to diagnosis: i) HRSD-24; or ii) Y-BOCS; or iii) BPRS | Change from baseline in HRSD-24 / Y-BOCS / BPRS at 2 months after final treatment
Score on rating scale that corresponds to diagnosis: i) HRSD-24; or ii) Y-BOCS; or iii) BPRS | Change from baseline in HRSD-24 / Y-BOCS / BPRS at 3 months after final treatment
Score on rating scale that corresponds to diagnosis: i) HRSD-24; or ii) Y-BOCS; or iii) BPRS | Change from baseline in HRSD-24 / Y-BOCS / BPRS at 6 months after final treatment

SECONDARY OUTCOMES:
Cognitive Functioning | Change from baseline in cognitive functioning at date of symptom remission or at date of 24th treatment, whichever comes first, assessed up to 12 weeks
  Improvement or sparing of cognitive functioning, as assessed by standard tests of episodic memory and non-memory cognitive functions.
Cognitive Functioning | Change from baseline in cognitive functioning at 6 months after final treatment
Neuroimaging (brain structure and activity) | Changes from baseline in brain structure and activity within 48 hours after final treatment
  Improvements in cortical thickness in subgenual cingulate cortex on T1 MRI voxel-based morphometry; improved anatomical connectivity between anterior hippocampus, subgenual cingulate cortex, and retrosplenial cortex on voxel-based comparative DTI tractography; subgenual and orbitofrontal functional connectivity to amygdala and ventral striatum on T2* fMRI BOLD signal covariation.
Neuroimaging (brain structure and activity) | Changes from baseline in brain structure and activity at 6 months after final treatment
  Improvements in cortical thickness in subgenual cingulate cortex on T1 MRI voxel-based morphometry; improved anatomical connectivity between anterior hippocampus, subgenual cingulate cortex, and retrosplenial cortex on voxel-based comparative DTI tractography; subgenual and orbitofrontal functional connectivity to amygdala and ventral striatum on T2* fMRI BOLD signal covariation.

CONTACTS AND LOCATIONS:
Overall Officials: Z. Jeffrey Daskalakis, MD, PhD., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Tang VM, Blumberger DM, Throop A, McClintock SM, Voineskos D, Downar J, Knyahnytska Y, Mulsant BH, Fitzgerald PB, Daskalakis ZJ. Continuation Magnetic Seizure Therapy for Treatment-Resistant Unipolar or Bipolar Depression. J Clin Psychiatry. 2021 Oct 19;82(6):20m13677. doi: 10.4088/JCP.20m13677. PMID 34670025
- [Derived] Weissman CR, Blumberger DM, Dimitrova J, Throop A, Voineskos D, Downar J, Mulsant BH, Rajji TK, Fitzgerald PB, Daskalakis ZJ. Magnetic Seizure Therapy for Suicidality in Treatment-Resistant Depression. JAMA Netw Open. 2020 Aug 3;3(8):e207434. doi: 10.1001/jamanetworkopen.2020.7434. PMID 32809030
- [Derived] Tang VM, Blumberger DM, Dimitrova J, Throop A, McClintock SM, Voineskos D, Downar J, Knyahnytska Y, Mulsant BH, Fitzgerald PB, Daskalakis ZJ. Magnetic seizure therapy is efficacious and well tolerated for treatment-resistant bipolar depression: an open-label clinical trial. J Psychiatry Neurosci. 2020 Sep 1;45(5):313-321. doi: 10.1503/jpn.190098. PMID 31922372
- [Derived] Tang VM, Blumberger DM, McClintock SM, Kaster TS, Rajji TK, Downar J, Fitzgerald PB, Daskalakis ZJ. Magnetic Seizure Therapy in Treatment-Resistant Schizophrenia: A Pilot Study. Front Psychiatry. 2018 Jan 16;8:310. doi: 10.3389/fpsyt.2017.00310. eCollection 2017. PMID 29387022
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.ca/en/research/Pages/research.aspx